CLINICAL TRIAL: NCT00907764
Title: An Open-Label, Parallel-Group, Exploratory Study to Evaluate the Efficacy and Safety of 400 ug Regadenoson Bolus for Pharmacological Stress Echocardiography
Brief Title: Stress Echocardiography Study With Regadenoson
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CVT 5127
Record Dates: First submitted 2009-05-20; First posted 2009-05-25 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Heart Disease; Coronary Artery Disease
MeSH Terms: conditions — Heart Diseases; Coronary Artery Disease | interventions — regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Regadenoson alone (Experimental)
  Interventions: Drug: regadenoson
- Regadenoson with exercise (Experimental)
  Interventions: Drug: regadenoson
- Regadenoson with contrast agent (Experimental)
  Interventions: Drug: regadenoson
- Regadenoson with contrast agent (perfusion) (Experimental)
  Interventions: Drug: regadenoson

INTERVENTIONS:
Drug: regadenoson — 400 ug, IV

SUMMARY:
Regadenoson is approved in the US under the brand name Lexiscan for myocardial perfusion imaging. This study will test whether regadenoson is an appropriate stress agent for stress echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinically indicated dobutamine echocardiogram showing normal wall motion at rest and abnormal wall motion with stress
* Patients with a clinically indicated dipyridamole echocardiogram showing normal perfusion and wall motion at rest and abnormal perfusion with or without abnormal wall motion with stress

Exclusion Criteria:

* Any condition precluding the safe administration of dobutamine, dipyridamole or SonoVue for echocardiography
* Pregnant or breast-feeding, or (if pre-menopausal), not practicing acceptable method of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Cardiac wall motion and perfusion abnormalities at rest and with regadenoson stress, with regadenoson stress and low level exercise, and with regadenoson stress and an echocontrast agent. | Within 12 minutes after dosing

SECONDARY OUTCOMES:
Various safety data will be collected, including adverse events, heart and blood pressure levels, ECG data, clinical laboratory results, and concomitant medications. | Up to day 29 after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Roxy Senior, Principal Investigator — Northwick Park Hospital
Locations (1):
- Northwick Park Hospital, Harrow, United Kingdom